CLINICAL TRIAL: NCT06452472
Title: Observational Study of People with Complete Hand Amputation Using a Multi-grip Myoelectric Prosthesis a Following Using a Standard Myoelectric Prosthesis
Acronym: PROMISE
Status: Completed | Type: Observational
Sponsor: Össur Iceland ehf (Industry)
Collaborators: Clin-Experts (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-A02856-49
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-06

CONDITIONS: Amputation of Upper Limb
Keywords: Amputation of upper limb; Observational Study; I-LIMB; multi-grip myoelectric hand prosthesis; function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: I-LIMB — Use of a multi-grip myoelectric hand prosthesis (I-LIMB after using a standard myoelectric prosthesis)

SUMMARY:
Cases of unilateral or bilateral upper limb amputation result in functional and aesthetic disability and a marked deterioration in quality of life. Amputees may use no prostheses, or use a combination of cosmetic prostheses, body-powered prostheses, or myoelectric prostheses (MHP). Among MHP, there are standard MHPs with a single degree of freedom (DOF) and one grip type, and multi-grip myoelectric hand (MG-MHP) with multiple DOF.

Amputees who do not use a prosthesis or a cosmetic prosthesis appear to have more difficulties in their daily activities and a greater disability than those who use body powered or myoelectric prostheses. While theoretically a MG-MHP offers the potential for subjects to perform more natural movements than a standard MHP, clinical evidence substantiating the advantages of MG-MHP over standard MHP in daily life remains inconclusive.

It remains essential to compare the advantages of MG-MHPs versus standard MHPs regarding functionality in daily life, quality of life and overall satisfaction among subjects who agree to transition from their standard MHP to a MG-MHP. The primary objective of this study was to assess upper limb function (specifically, the upper limb function component of the Orthotics and Prosthetics Users' Survey (OPUS) questionnaire) provided by a specific MG-MHP, i-Limb®, compared to a standard MHP in subjects with complete hand amputation.

The subjects participating in the study were patients equipped with MHP, coming to the center for a MG-MHPs hand test. If the prescription for the MG-MHPs hand was validated, the patient was then followed in the study for 8 to 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years old
* Patient with a unilateral acquired or congenital complete amputation
* Patient using a standard myoelectric hand prosthesis for at least 4 weeks
* Patient who has an indication of a Multi-Grip Myoelectric Hand Prosthesis , according to a multidisciplinary team

Exclusion Criteria:

* Pregnant women
* Patient under guardianship
* Patient with multiple amputations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators involved in the study are all doctors specializing in the fitting of limb amputee subjects. The study is conducted in French physical medicine and rehabilitation centers.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Change in daily living with his/her prosthesis | at 8-10 weeks
  Assessed with upper limb function component of the Orthotics and prosthetics Users 'Survey (OPUS) which includes 23 questions and explores the ease with which the subject performs 23 activities of daily living with his/her prosthesis. The questions are rated from 4 very easy; 3 Easy 2 Slightly difficult; 1 Very difficult; 0 Cannot perform activity. The total score ranges from a minimum of 0 to a maximum of 92. A higher score correlates with an enhanced perception of functional

SECONDARY OUTCOMES:
Change in the quality-of-life with his/her prosthesis | at 8-10 weeks
  Assessed with the OPUS quality of life score which includes 23 questions rated in 5 points. Questions 1 to 12 explore the subject's feelings on 12 aspects of their quality of life and interpersonal relationships, which are rated for overall feeling as follows: 4 None of the time; 3 A little of the time; 2 Some of the time ; 1 Most of the time ; 0 All the time. Questions 13 to 23 explore the subject's feelings about 11 aspects of their quality of life in terms of psychological experience and are rated as follow 4 all the time;3 Most of the time; 2 Some of the time; 1 A little of the time; 0 None of the time The total score is a minimum of 0 and a maximum of 92. The higher the score, the better the subject's quality of life
Change is the satisfaction of the patient with his/her prosthesis | at 8-10 weeks
  Assessed with the prosthesis satisfaction dimension of the OPUS which includes 11 questions which explores 11 characteristics about the prosthesis. The questions are rated as follow: questions are rated as follows: 5 Strongly agree; 4 Agree; 3 Neither agree nor disagree : 2 Disagree; 1 Strongly disagree. The subject can answer "don't know". The total score is a minimum of 11 and a maximum of 55. The higher the score, the greater the subject's satisfaction with their prosthesis.
Change is the satisfaction of the patient to the services provided assessed with OPUS | at 8-10 weeks
  Assessed with the satisfaction dimension relating to the services of the OPUS explores 10 characteristics associated with the services connected to the utilization of the prosthesis.. Questions are rated as follows: 5 Strongly agree; 4 Agree; 3 neither agree nor disagree; 2 Disagree; 1 Strongly disagree. The total score is a minimum of 10 and a maximum of 50. The higher the score, the greater the subject's satisfaction with their prosthesis
Change in satisfaction of the patient assessed with ESAT | at 8-10 weeks
  Assess the change in satisfaction of the patient with Quebec User Evaluation of Satisfaction with assistive Technology (QUEST = ESAT in French); A higher score indicates higher satisfaction
Change in the Quick-DASH functional scale | at 8-10 weeks
  The Quick DASH is an 11-item questionnaire designed to assess symptoms and functional limitations in individuals with upper limb disorders . It provides a 100% summative score, with 100 indicating the greatest handicap.
Change in the overall satisfaction of the patient on a Likert scale | at 8-10 weeks
  Overall satisfaction on an 11-point Likert scale rated from 0 (not at all satisfied) to 10 (totally satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle LOIRET, MD, Principal Investigator — IRR - Établissement de Nancy - Louis-Pierquin
Locations (1):
- Multiples Facilities, Multiple Locations, France

IPD SHARING:
Plan to Share IPD: No